CLINICAL TRIAL: NCT01397903
Title: A Cross-sectional Observational Study to Describe Treatment Management of Patients With Major Depressive Disorder (MDD) and Inadequate Response to Antidepressants in Greece
Brief Title: Description of Treatment Management of Patients With Major Depressive Disorder and Inadequate Response
Acronym: MADDRE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-NGR-XXX-2011/1
Record Dates: First submitted 2011-07-18; First posted 2011-07-20 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Major Depressive Disorder
Keywords: antidepressant therapy, inadequate control, add-on therapy
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Group 1: Inpatients and outpatients diagnosed with major depressive disorder as per the DSM-IV criteria who had poor disease control during antidepressant treatment and have completed 4 weeks of add-on drug therapy at enrolment in the study.
  The percentage of patients with CGI-I score ≤ 2 at study Visit (4 weeks after the commencement of add-on treatment).

SUMMARY:
The purpose is to assess the response of add-on therapy, based on CGI-I scale, at 4 weeks, in patients with MDD who had an inadequate disease control with antidepressant medication.

DETAILED DESCRIPTION:
A cross-sectional observational study to describe treatment management of patients with Major Depressive Disorder (MDD) and inadequate response to antidepressants in Greece

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MDD as per DSM-IV
* Patients with an inadequate disease control during antidepressant therapy
* Patients who already receive add-on therapy and have completed 4-5 weeks of treatment at the time of their enrolment in the study.

Exclusion Criteria:

* Patients fulfilling criteria for diagnosis of any other psychiatric condition (except for MDD), as per DSM-IV Axis I,
* Concomitant organic mental disorder or mental retardation Substance abuse or dependence (with the exception of nicotine dependence), as defined by DSM-IV criteria Participation in another study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Psychiatric patients
Sampling Method: Probability Sample
Enrollment: 545 (Actual)
Dates: Start 2011-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
To assess the response of additional therapy by assessment of percentage of patients with CGI-I score ≤ 2 | At week 4 after the commencement of add-on therapy

SECONDARY OUTCOMES:
Number of consecutive treatments administered for the management of the current MDD episode until the commencement of adjunctive (add-on) medication. | At week 4 after the commencement of add-on therapy
Percentage of patients (n, %) with MADRS score ≤ 10 at week 4 following the onset of adjunctive medication | At week 4 following the onset of add-on medication
Percentage of patients (n,%) with a change (decrease) in MADRS score be ≥ 50% | At week 4 following the initiation of add-on drug therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Pontikis, Study Director — Marketing Company Medical and Regulatory Affairs Director, AstraZeneca S.A. Greece
Locations (27):
- Greece (27):
  - Research Site, Arta, Artas
  - Research Site, Athens, Attica
  - Research Site, Chaïdári, Attica
  - Research Site, Dafni, Attica
  - Research Site, Glyfada, Attica
  - Research Site, Kifissia, Attica
  - Research Site, Koropí, Attica
  - Research Site, Marousi, Attica
  - Research Site, Nea Makri, Attica
  - Research Site, Peristeri, Attica
  - Research Site, Petroúpolis, Attica
  - Research Site, Rhodes, Dodekanese
  - Research Site, Agrinio, Etoloacarnania
  - Research Site, Lamia, Fhiotida
  - Research Site, Heraklio, Heraklio
  - Research Site, Ioannina, Ioanninon
  - Research Site, Kalamata, Kalamata
  - Research Site, Karditsa, Karditsa
  - Research Site, Kavala, Kavala
  - Research Site, Larissa, Larissa
  - Research Site, Ag. Nikolaos, Lasithiou
  - Research Site, Pátrai, Patras
  - Research Site, Aigáleo, Piraeus
  - Research Site, Serres, Serres
  - Research Site, Thessaloniki, Thessaloniki
  - Research Site, Trikala, Trikala
  - Research Site, Thebes, Viotia